CLINICAL TRIAL: NCT06903546
Title: The Effect of Propolis Administration on Low Density Lipoprotein and High Density Lipoprotein in Diabetic Type 2 Patients in Central Jakarta
Brief Title: The Effect of Propolis Administration on Cholesterol Level in Diabetic Type 2 Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. drg. Dwirini Retno Gunarti, M.S., Associate Professor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 24-10-1677
Record Dates: First submitted 2025-03-28; First posted 2025-03-30 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Propolis; Diabetes Mellitus Type 2; Low Density Lipoprotein; High Density Lipoprotein
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated into two groups that will recieve either propolis or plasebo. The study model is double-blinded trial.
  The participants are patients undergoing treatment for type 2 diabetes in multiple sub-dictrict health centre in Central Jakarta and will be screened based on inclusion and exclusion criteria.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): This group will receive the intervention, which in this study is propolis with dose given 1 drop/kg/time given, 2 times daily, for 8 weeks (2 months)
  Interventions: Drug: Propolis drops
- Control group (Placebo Comparator): This group will receive placebo (a look-alike substance that contains no drug) with dose given 1 drop/kg/time given, 2 times daily, for 8 weeks (2 months)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Propolis drops — The intervention given is propolis drops that are approved by Indonesian Food and Drug Authority
  Arms: Intervention group
Other: Placebo — The given placebo are look-alike substance with no effect
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if propolis administration works to change the level of Low Density Lipoprotein (LDL) and High Density Lipoprotein cholesterol (HDL) in diabetic type 2 patients.

The main questions it aims to answer are:

- Is giving 1 drops/ 10kg/ times, twice daily for 8 weeks will change the level of LDL and HDL level in diabetic type 2 patients compared to placebo? Researchers will compare propolis to a placebo (a look-alike substance that contains no drug) to see if propolis works to change LDL and HDL cholesterol level.

Participants will:

* Take propolis or a placebo, 2 times daily with given dose (1 drops/10 kg/times) every day for 2 months
* Visit the sub-district health centre once every 2 weeks for checkups
* Get their blood checked before and after intervention

DETAILED DESCRIPTION:
Subject allocation into groups will be made by third party to ensure masking/ blinding protocol.

Data that will be taken from participants :

* Private information
* Medication history (for type 2 Diabetes Mellitus)
* Food intake (calories, fats, carbohydrate, protein, and flavonoid intake)
* Physical activity status

ELIGIBILITY:
Inclusion Criteria:

* Controlled Diabetes Mellitus type 2 with HbA1c <7.5%
* BMI 23-35 kg/m2
* On anti-cholesterol therapy

Exclusion Criteria:

* Using injection therapy (insulin or GLP-1 RA)
* History of bees product allergy
* Active smoker
* Consuming alcohol
* Altered liver (ALT>35 IU/L) and kidney (eGFR<90 mL/min) function
* Pregnant and breastfeeding women
* History of cardiovascular disease (heart attack, stroke)

Ages: 35 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male and female
Enrollment: 64 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Low Density Lipoprotein | 8 weeks
  LDL level will be measured twice, before and after intervention
High Density Lipoprotein | 8 weeks
  HDL will be measured twice, before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dwirini R Gunarti, Biomed Science, Principal Investigator — Indonesia University
Locations (1):
- University of Indonesia Faculty of Biomedical Science, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
Confidentiality issue

REFERENCES:
- [Background] Zakerkish M, Jenabi M, Zaeemzadeh N, Hemmati AA, Neisi N. The Effect of Iranian Propolis on Glucose Metabolism, Lipid Profile, Insulin Resistance, Renal Function and Inflammatory Biomarkers in Patients with Type 2 Diabetes Mellitus: A Randomized Double-Blind Clinical Trial. Sci Rep. 2019 May 13;9(1):7289. doi: 10.1038/s41598-019-43838-8. PMID 31086222
- [Background] Samadi N, Mozaffari-Khosravi H, Rahmanian M, Askarishahi M. Effects of bee propolis supplementation on glycemic control, lipid profile and insulin resistance indices in patients with type 2 diabetes: a randomized, double-blind clinical trial. J Integr Med. 2017 Mar;15(2):124-134. doi: 10.1016/S2095-4964(17)60315-7. PMID 28285617